CLINICAL TRIAL: NCT02695615
Title: The Evaluation of the Effects of Stress During Elective or Emergency Cesarean Operations; Prospective, Randomized Clinical Trial
Brief Title: Stress During Elective or Emergency Cesarean Operations
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gulsah Karaoren, MD, Umraniye Education and Research Hospital
Other Study IDs: GK10
Record Dates: First submitted 2016-02-24; First posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Anxiety
Keywords: cesarean operation; Spielberger State Trait Anxiety Inventory; pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
We investigated a correlation between maternal anxiety and age, body mass index (BMI), parity-gravidity, patient satisfaction, antenatal care, postoperative pain according to emergent or elective C/S under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women aged ≥18 years (gestational age: 37-40 weeks) underwent emergent or elective C/S.

Exclusion Criteria:

* patients with cardiopulmonary,
* renal,
* hepatic or
* psychiatric disease,
* obstetric-fetal anomaly and
* weighing ≥ 100 kg were excluded.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study included pregnant women aged ≥18 years (gestational age: 37-40 weeks) in whom emergent or elective C/S was indicated
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
correlation between maternal anxiety and age according to emergent or elective C/S under general anesthesia. | during operation
correlation between maternal anxiety and body mass index according to emergent or elective C/S under general anesthesia. | during operation

SECONDARY OUTCOMES:
correlation between maternal anxiety and parity-gravidity according to emergent or elective C/S under general anesthesia. | during the operation
correlation between maternal anxiety and patient satisfaction according to emergent or elective C/S under general anesthesia. | during the operation
correlation between maternal anxiety and postoperative pain according to emergent or elective C/S under general anesthesia. | during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed A Erkmen, MD, Study Chair — Umraniye Education and Research Hospital
Locations (1):
- gulsah Karaoren, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duggan M, Dowd N, O'Mara D, Harmon D, Tormey W, Cunningham AJ. Benzodiazepine premedication may attenuate the stress response in daycase anesthesia: a pilot study. Can J Anaesth. 2002 Nov;49(9):932-5. doi: 10.1007/BF03016877. PMID 12419719